CLINICAL TRIAL: NCT03932994
Title: Development and Evaluation of ACT on Health: An Online Health Promotion Program
Brief Title: Evaluation of the ACT on Health Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Levin, Associate Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOH2018
Record Dates: First submitted 2019-04-15; First posted 2019-05-01 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT on Health Intervention (Experimental): Those assigned to ACT on Health will use the program over the next 8 weeks, completing weekly modules and coaching calls.
  Interventions: Behavioral: ACT on Health
- Waitlist (No Intervention): Those assigned to the waitlist will simply wait 8 weeks. A second online assessment will be completed 8 weeks after baseline in both conditions (for a between condition comparison). After the second assessment, waitlist participants will gain access to ACT on Health.

INTERVENTIONS:
Behavioral: ACT on Health — This intervention consists of an online canvas course based on Acceptance and Commitment Therapy, focused on increasing healthy diet and physical activity and addressing barriers to change. The intervention also consists of weekly phone coaching calls.
  Arms: ACT on Health Intervention

SUMMARY:
This project will develop and test an online health promotion program that augments diet and physical activity behavior change methods using acceptance and commitment therapy (ACT). ACT is an evidence-based cognitive behavioral therapy found to be effective in over 200 randomized controlled trials (RCTs) in improving a wide range of psychological and behavioral health problems. Recently, several clinical trials have found ACT enhances diet and exercise behavior as well as long term weight management. These studies have focused on testing ACT provided by experts in face-to-face interventions, which limits broad dissemination. Delivering an ACT health promotion program online could potentially provide a low-cost resource to improve health across Utah.

The specific aims are to:

1. Develop a canvas-based online course (ACT on Health) that teaches how to improve diet and physical activity as well as ACT-based skills to enhance behavior change efforts.
2. Evaluate ACT on Health relative to a waitlist in a RCT with 60 overweight/obese adults on outcomes including self-reported physical activity, diet, and quality of life.

If successful, this project will both provide an ongoing canvas extension course delivered throughout Utah to improve health behaviors.

This project seeks to develop and test an online, self-guided ACT program (ACT on Health) to improve diet and physical activity. ACT on Health will include 8 weekly modules teaching effective health behavior change methods coupled with ACT strategies to reduce maladaptive motivators and enhance adaptive motivators for change. The investigators will evaluate the program in a RCT relative to a waitlist condition with 60 overweight/obese adults recruited through Extension in 7 Utah counties. The program will be offered through the USU Extension Canvas platform to ensure, if effective, that the program could continue to be offered across Utah.

The two hypotheses for this study are as follows:

1. Participants will report a high degree of satisfaction and will demonstrate adequate engagement in the ACT on Health program.
2. Participants assigned to ACT on Health will improve more on self-reported diet, physical activity, and quality of life relative to the waitlist condition.

DETAILED DESCRIPTION:
This project will develop and test an online health promotion program that augments diet and physical activity behavior change methods using acceptance and commitment therapy (ACT). ACT is an evidence-based cognitive behavioral therapy found to be effective in over 200 randomized controlled trials (RCTs) in improving a wide range of psychological and behavioral health problems. Recently, several clinical trials have found ACT enhances diet and exercise behavior as well as long term weight management. These studies have focused on testing ACT provided by experts in face-to-face interventions, which limits broad dissemination. Delivering an ACT health promotion program online could potentially provide a low-cost resource to improve health across Utah. The specific aims are to:

1. Develop a canvas-based online course (ACT on Health) that teaches how to improve diet and physical activity as well as ACT-based skills to enhance behavior change efforts.
2. Evaluate ACT on Health relative to a waitlist in a RCT with 60 overweight/obese adults on outcomes including self-reported physical activity, diet, and quality of life.

If successful, this project will both provide an ongoing canvas extension course delivered throughout Utah to improve health behaviors.

Background and Significance Obesity and its contributing behaviors (i.e., physical inactivity, poor diet) are significant public health issues. Obesity is associated with a range of serious medical conditions, decreased life expectancy, and impaired quality of life. Physical inactivity contributes to premature mortality and cardiovascular disease above and beyond its impact on obesity. In contrast, healthy diet and exercise decreases risk for a wide range of medical conditions and premature mortality. Epidemiological research indicates 69% of US adults are obese or overweight. Furthermore, only 23% of adults meet recommended guidelines for physical activity, and only 24% of adults eat five or more serving of fruits and vegetables per day. The prevalence of obesity and poor health behaviors, despite their negative consequences, highlight how difficult it is to make sustained changes to health behaviors.

Motivation is a key factor for improving and maintaining healthy diet and physical activity. There is a substantial literature on the importance of intrinsic motivation for health behavior change, in which individuals are personally motivated for positive reasons inherent to them or the activity (e.g., enjoyment, values). For example, intrinsic motivation predicts healthier exercise and diet and improvements in intrinsic motivation mediate obesity intervention effects.

In addition to a lack of intrinsic motivation, individuals who are overweight often struggle with an excess of controlled motivators for behavior change based on a sense of "having to" act to avoid negative consequences or feelings. In contrast to intrinsic motivation, greater controlled motivation predicts poorer diet, physical inactivity, and quality of life. These challenges are exacerbated by the prevalent stigma obese people encounter in daily life. Internalizing stigmatizing attitudes (i.e., weight self-stigma) can drive controlled motivators for weight loss out of fear of being stigmatized by others (e.g. "so people don't make fun of me") or devaluing oneself (e.g., "because I'm so ashamed of myself"), which overshadow effective, intrinsic motivators. As a result, weight self-stigma can lead to exercise avoidance, unhealthy eating, lower adherence to weight loss programs, and worse health outcomes.

Currently there is a lack of interventions targeting both maladaptive, controlled motivators (particularly those resulting from internalizing stigmatizing messages about weight), in addition to adaptive, intrinsic motivators for behavior change. Innovative interventions are needed that can improve obesity and associated health behaviors by increasing intrinsic motivation, while decreasing problematic motivators (e.g., shame, self-judgment, external pressure) that impede meaningful, sustained behavior change.

Acceptance and commitment therapy (ACT) is one promising approach for addressing such motivational factors in health behavior change. ACT uses acceptance and mindfulness based strategies to target maladaptive motivators, and values and commitment strategies to increase intrinsic motivation for change. Through these strategies, ACT teaches people how to change behavior to move towards what matters, in a compassionate, meaningful way. ACT was originally developed for problems such as depression and anxiety, which is why it has developed such robust methods for addressing psychological barriers. Fortunately, it has been expanded to treat behavioral health issues as well. To-date 14 RCTs have evaluated ACT for weight management or physical activity, finding ACT improves physical activity, healthy eating, and weight loss relative to waitlist, treatment as usual, and in some cases, standard behavioral weight loss programs. ACT has also been found to improve stigma and health behaviors among those struggling with weight self-stigma.

ACT weight management research has primarily focused on expert delivered, intensive face- to-face programs, as long as 37 hours of groups over 40 weeks. Such programs stem from challenges with obtaining sustained, meaningful weight loss. However, these programs are burdensome to participate in, resource intensive to deliver, and require a local expert provider. This translates into less reach to those in need; particularly individuals with less availability, resources, or opportunities to participate in intensive face-to-face ACT.

Online self-guided programs can address many of these barriers. A self-paced online ACT program allows participation irrespective of location or schedule, and at a low cost that can translate into sustainable, large-scale community interventions. The investigator's research has found ACT can be effectively delivered online to treat mental health concerns in six published clinical trials. Of more direct relevance, the investigators completed two small pilot trials in which self-guided ACT interventions improved diet and physical activity through targeting weight self-stigma and intrinsic motivation. These results suggest a comprehensive online ACT program that targets both maladaptive motivators related to weight self-stigma and increases adaptive motivators for health behavior change could provide an effective, far reaching program to improve public health.

This project seeks to develop and test an online, self-guided ACT program (ACT on Health) to improve diet and physical activity. ACT on Health will include 8 weekly modules teaching effective health behavior change methods coupled with ACT strategies to reduce maladaptive motivators and enhance adaptive motivators for change. The investigators will evaluate the program in a RCT relative to a waitlist condition with 60 overweight/obese adults recruited through Extension in 7 Utah counties. The program will be offered through the USU Extension Canvas platform to ensure, if effective, that the program could continue to be offered across Utah.

Approach Project timeline and objectives. The objectives of this project are to 1) develop a canvas- based online course (ACT on Health), and 2) evaluate ACT on Health in a RCT.

ACT on Health Program. The program will include 8 weekly modules completed in an asynchronous format (i.e., register and start any time). Each module will include a combination of text, video lectures, audio-guided exercises, and interactive worksheets. The weekly modules will build upon each other, covering key methods for enhancing diet and physical activity as well as ACT strategies to address motivation and related barriers (e.g., weight self-stigma, cognitive and affective barriers). Participants will set a weekly goal related to the new skills they learned. To support program adherence, phone coaching calls will be provided weekly by a graduate student in the clinical/counseling psychology Ph.D. program. Calls will be 5-10 minutes long and based on the investigator's protocol from a self-help book study for weight self-stigma. ACT on Health will be developed on Canvas. Dr. Levin has over 10 years of experience creating online ACT courses using similar platforms, which provide an efficient, effective way to develop an engaging program. Content related to diet and physical activity will be developed by Dr. Durward and extension faculty, who have extensive expertise in this area, while content related to ACT will be developed by Dr. Levin. Content will be developed iteratively, obtaining feedback on drafts from the research team, and translating it to a final online course.

Evaluation Plan Participants and Recruitment. The investigators will evaluate ACT on Health relative to a waitlist in a RCT with 60 overweight/obese adults. Eligibility criteria include being 18 or older, a self-reported body mass index of 25 or higher, and interested in participating in an online program to improve eating and physical activity. No other exclusion criteria will be used in order to ensure a representative sample and to maximize participant flow. The investigators will recommend participants consult their physician if they have a condition that might be affected by changes to diet or exercise.

Extension faculty will recruit potential participants across 7 Utah counties. Recruitment flyers will be posted in local community areas and events (e.g., grocery stores, coffee shops, libraries, farmers' markets), sent out through email lists, and posted online on community websites. Local providers (e.g., doctor's offices, dietitians) will also be asked to distribute flyers.

Procedures. Participants will complete all study procedures online and through phone calls. Participants will first complete an online screening, consent, and then baseline assessment delivered through Qualtrics. After completing the baseline assessment, participants will be automatically randomized to either the ACT on Health or waitlist condition.

Those assigned to ACT on Health will use the program over the next 8 weeks, completing weekly modules and coaching calls. Those assigned to the waitlist will simply wait 8 weeks. A second online assessment will be completed 8 weeks after baseline in both conditions (for a between condition comparison). After the second assessment, waitlist participants will gain access to ACT on Health. A third online assessment will be completed 8 weeks later (16 weeks after baseline), providing a within condition follow up assessment for the intervention condition and a within condition pre-post replication for the waitlist condition (whether waitlisted participants who began using ACT on Health at week 8 demonstrated improvements at week 16).

ELIGIBILITY:
Inclusion Criteria:

* Being 18 or older.
* Being a fluent English speaker.
* A self-reported body mass index of 25 or higher.
* Interest participating in an online program to improve eating and physical activity.
* Regular access to the internet.
* Comfort with using the internet and navigating websites.
* Living in Utah or neighboring counties.
* Have not participated in other web/mobile or self-help book studies from the USU CBS lab.

Exclusion Criteria:

* No other exclusion criteria will be used in order to ensure a representative sample and to maximize participant flow
* We will recommend participants consult their physician if they have a condition that might be affected by changes to diet or exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Automated Self-Administered 24-hour Dietary Assessment Tool (ASA24) | 24 hours
  Asks participants to report on the specific foods they ate over the past day to measure specific nutritional intake

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 1 week
  Measures types and length of physical activity performed in the last week. The questionnaire can be scored using the number of minutes spent doing physical activity or by categorizing into low (less physical activity reported than the specified amounts for medium or high physical activity), medium (at least half an hour of at least moderate physical activity on most days), and high physical activity (1 hour or more of at least moderate physical activity per day).
Three Factor Eating Questionnaire (TFEQ) | 8 weeks
  Measures dietary restraint, disinhibited eating, and predisposition to hunger. The TFEQ has three subscales: dietary restraint (ranging from 0-21), disinhibition (ranging from 0-16), and hunger (ranging from 0-14). Greater scores indicate greater dietary restraint, disinhibition, and hunger.
Weight Control Strategies Scale (WCSS) | 8 weeks
  Measures use of specific behaviors thought to help weight loss. This scale has four subscales: Dietary Choices (10 items, ranging from 0-40), Self-monitoring Strategies (7 items, ranging from 0-28), Physical Activity (6 items, ranging from 0-24), and Psychological Coping (7 items, ranging from 0-28). The total score can range from 0-120. Scores are established by adding up all items. Greater scores mean greater use of weight control strategies as specified by the subscales.
General Health Questionnaire (GHQ) General Health Questionnaire | 2 weeks
  Measure of psychological morbidity and general distress. The total score can range from 12-28, with higher scores indicating greater psychological health.
Weight Self Stigma Questionnaire (WSSQ) | During the past month
  Measures self-devaluation and fear of enacted stigma in overweight individuals. There are two subscales, self-devaluation and fear of enacted stigma, added together to form the total score. The total scores range from 12-60, with higher scores indicating greater weight self stigma. The subscale scores both range from 6-30 with higher scores indicating greater self-devaluation and fear of enacted stigma.
Acceptance and Action Questionnaire for Weight-Related Difficulties (AAQ-W) | 8 weeks
  Measures experiential avoidance of weight-related thoughts, feelings, and experiences.

CONTACTS AND LOCATIONS:
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: No